CLINICAL TRIAL: NCT00557193
Title: A Phase III Study of Risk Directed Therapy for Infants With Acute Lymphoblastic Leukemia (ALL): Randomization of Highest Risk Infants to Intensive Chemotherapy +/- FLT3 Inhibition (CEP-701, Lestaurtinib; NSC#617807)
Brief Title: Combination Chemotherapy With or Without Lestaurtinib in Treating Younger Patients With Newly Diagnosed Acute Lymphoblastic Leukemia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Children's Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AALL0631; NCI-2009-00313 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CDR0000573996; 08-146; COG-AALL0631; AALL0631 (Other: Children's Oncology Group); AALL0631 (Other: CTEP); U10CA098543 (NIH); U10CA180886 (NIH)
Record Dates: First submitted 2007-11-09; First posted 2007-11-12 (Estimated); Results first posted 2018-12-10 (Actual); Last update posted 2024-07-15 (Actual); Status verified 2024-07

CONDITIONS: Acute Lymphoblastic Leukemia; Acute Undifferentiated Leukemia; Childhood T Acute Lymphoblastic Leukemia
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma; Leukemia, Biphenotypic, Acute | interventions — Asparaginase; Leyk; Specimen Handling; Biopsy; Cyclophosphamide; Cytarabine; Daunorubicin; Dexamethasone; Calcium Dobesilate; auricularum; dexamethasone acetate; dexamethasone 21-phosphate; Etoposide; Filgrastim; Granulocyte Colony-Stimulating Factor; lestaurtinib; Leucovorin; Mercaptopurine; azathiopurine; Methotrexate; merphos; Methylprednisolone; exifone; Medrol Veriderm; pegaspargase; Prednisone; deltacortene; prednylidene; Hydrocortisone; Vincristine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Arm A (standard risk MLL-G) (Experimental): Population Description: Eligible patients with MLL-G (germline, or non-rearranged)
  Interventions: Drug: Asparaginase; Procedure: Biospecimen Collection; Procedure: Bone Marrow Biopsy; Drug: Cyclophosphamide; Drug: Cytarabine; Drug: Daunorubicin Hydrochloride; Drug: Dexamethasone; Procedure: Echocardiography; Drug: Etoposide; Biological: Filgrastim; Other: Laboratory Biomarker Analysis; Drug: Leucovorin Calcium; Drug: Mercaptopurine; Drug: Methotrexate; Drug: Methylprednisolone; Procedure: Multigated Acquisition Scan; Drug: Pegaspargase; Other: Pharmacological Study; Drug: Prednisone; Drug: Therapeutic Hydrocortisone; Drug: Vincristine Sulfate
- Arm B (IR/HR MLL-R chemotherapy) (Active Comparator): Population Description: Eligible patients with MLL-R (rearranged). Considered Intermediate Risk (IR) if age >= 90 days at diagnosis and High Risk (HR) if age < 90 days at diagnosis.
  Interventions: Drug: Asparaginase; Procedure: Biospecimen Collection; Procedure: Bone Marrow Biopsy; Drug: Cyclophosphamide; Drug: Cytarabine; Drug: Daunorubicin Hydrochloride; Drug: Dexamethasone; Procedure: Echocardiography; Drug: Etoposide; Biological: Filgrastim; Other: Laboratory Biomarker Analysis; Drug: Leucovorin Calcium; Drug: Mercaptopurine; Drug: Methotrexate; Drug: Methylprednisolone; Procedure: Multigated Acquisition Scan; Drug: Pegaspargase; Other: Pharmacological Study; Drug: Prednisone; Drug: Therapeutic Hydrocortisone; Drug: Vincristine Sulfate
- Arm C (IR/HR MLL-R chemotherapy and lestaurtinib) (Experimental): Population Description: Eligible patients with MLL-R (rearranged). Considered Intermediate Risk (IR) if age >= 90 days at diagnosis and High Risk (HR) if age < 90 days at diagnosis.
  Interventions: Drug: Asparaginase; Procedure: Biospecimen Collection; Procedure: Bone Marrow Biopsy; Drug: Cyclophosphamide; Drug: Cytarabine; Drug: Daunorubicin Hydrochloride; Drug: Dexamethasone; Procedure: Echocardiography; Drug: Etoposide; Biological: Filgrastim; Other: Laboratory Biomarker Analysis; Drug: Lestaurtinib; Drug: Leucovorin Calcium; Drug: Mercaptopurine; Drug: Methotrexate; Drug: Methylprednisolone; Procedure: Multigated Acquisition Scan; Drug: Pegaspargase; Other: Pharmacological Study; Drug: Prednisone; Drug: Therapeutic Hydrocortisone; Drug: Vincristine Sulfate

INTERVENTIONS:
Drug: Asparaginase — Given IV, IM, or PO
  Other Names: ASP-1; Asparaginase II; Asparaginase-E.Coli; Colaspase; Elspar; Kidrolase; L-Asnase; L-ASP; L-Asparaginase; L-Asparagine Amidohydrolase; Laspar; Lcf-ASP; Leucogen; Leunase; MK-965; Paronal; Re-82-TAD-15; Serasa; Spectrila
Procedure: Biospecimen Collection — Undergo blood sample collection
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Procedure: Bone Marrow Biopsy — Undergo bone marrow biopsy
  Other Names: Biopsy of Bone Marrow; Biopsy, Bone Marrow
Drug: Cyclophosphamide — Given IV
  Other Names: (-)-Cyclophosphamide; 2H-1,3,2-Oxazaphosphorine, 2-[bis(2-chloroethyl)amino]tetrahydro-, 2-oxide, monohydrate; Asta B 518; B 518; B-518; B518; Carloxan; Ciclofosfamida; Ciclofosfamide; Cicloxal; Clafen; Claphene; CP monohydrate; CTX; CYCLO-cell; Cycloblastin; Cycloblastine; Cyclophospham; Cyclophosphamid monohydrate; Cyclophosphamide Monohydrate; Cyclophosphamidum; Cyclophosphan; Cyclophosphane; Cyclophosphanum; Cyclostin; Cyclostine; Cytophosphan; Cytophosphane; Cytoxan; Fosfaseron; Genoxal; Genuxal; Ledoxina; Mitoxan; Neosar; Revimmune; Syklofosfamid; WR 138719; WR- 138719; WR-138719; WR138719
Drug: Cytarabine — Given IV or IT
  Other Names: .beta.-Cytosine arabinoside; 1-.beta.-D-Arabinofuranosyl-4-amino-2(1H)pyrimidinone; 1-.beta.-D-Arabinofuranosylcytosine; 1-Beta-D-arabinofuranosyl-4-amino-2(1H)pyrimidinone; 1-Beta-D-arabinofuranosylcytosine; 1.beta.-D-Arabinofuranosylcytosine; 2(1H)-Pyrimidinone, 4-Amino-1-beta-D-arabinofuranosyl-; 2(1H)-Pyrimidinone, 4-amino-1.beta.-D-arabinofuranosyl-; Alexan; Ara-C; ARA-cell; Arabine; Arabinofuranosylcytosine; Arabinosylcytosine; Aracytidine; Aracytin; Aracytine; Beta-Cytosine Arabinoside; CHX-3311; Cytarabinum; Cytarbel; Cytosar; Cytosine Arabinoside; Cytosine-.beta.-arabinoside; Cytosine-beta-arabinoside; Erpalfa; Starasid; Tarabine PFS; U 19920; U-19920; Udicil; WR-28453
Drug: Daunorubicin Hydrochloride — Given IV
  Other Names: Cerubidin; Cerubidine; Cloridrato de Daunorubicina; Daunoblastin; Daunoblastina; Daunoblastine; Daunomycin Hydrochloride; Daunomycin, hydrochloride; Daunorubicin.HCl; Daunorubicini Hydrochloridum; FI-6339; Ondena; RP-13057; Rubidomycin Hydrochloride; Rubilem
Drug: Dexamethasone — Given IV or PO
  Other Names: Aacidexam; Adexone; Aknichthol Dexa; Alba-Dex; Alin; Alin Depot; Alin Oftalmico; Amplidermis; Anemul mono; Auricularum; Auxiloson; Baycadron; Baycuten; Baycuten N; Cortidexason; Cortisumman; Decacort; Decadrol; Decadron; Decadron DP; Decalix; Decameth; Decasone R.p.; Dectancyl; Dekacort; Deltafluorene; Deronil; Desamethasone; Desameton; Dexa-Mamallet; Dexa-Rhinosan; Dexa-Scheroson; Dexa-sine; Dexacortal; Dexacortin; Dexafarma; Dexafluorene; Dexalocal; Dexamecortin; Dexameth; Dexamethasone Intensol; Dexamethasonum; Dexamonozon; Dexapos; Dexinoral; Dexone; Dinormon; Dxevo; Fluorodelta; Fortecortin; Gammacorten; Hemady; Hexadecadrol; Hexadrol; LenaDex; Lokalison-F; Loverine; Methylfluorprednisolone; Millicorten; Mymethasone; Orgadrone; Spersadex; TaperDex; Visumetazone; ZoDex
Procedure: Echocardiography — Undergo ECHO
  Other Names: EC
Drug: Etoposide — Given IV
  Other Names: Demethyl Epipodophyllotoxin Ethylidine Glucoside; EPEG; Lastet; Toposar; Vepesid; VP 16; VP 16-213; VP 16213; VP-16; VP-16-213; VP-16213; VP16; VP16213
Biological: Filgrastim — Given IV or SC
  Other Names: Filgrastim Biosimilar Filgrastim-sndz; Filgrastim Biosimilar Tbo-filgrastim; Filgrastim XM02; Filgrastim-aafi; Filgrastim-ayow; Filgrastim-sndz; G-CSF; Granix; Neupogen; Neutroval; Nivestim; Nivestym; r-metHuG-CSF; Recombinant Methionyl Human Granulocyte Colony Stimulating Factor; Releuko; rG-CSF; Tbo-filgrastim; Tevagrastim; XM02; Zarxio
Other: Laboratory Biomarker Analysis — Correlative studies
Drug: Lestaurtinib — Given PO
  Other Names: CEP 701; CEP-701; CEP701; KT-5555; SPM-924
  Arms: Arm C (IR/HR MLL-R chemotherapy and lestaurtinib)
Drug: Leucovorin Calcium — Given IV
  Other Names: Adinepar; Calcifolin; Calcium (6S)-Folinate; Calcium Folinate; Calcium Leucovorin; Calfolex; Calinat; Cehafolin; Citofolin; Citrec; Citrovorum Factor; Cromatonbic Folinico; Dalisol; Disintox; Divical; Ecofol; Emovis; Factor, Citrovorum; Flynoken A; Folaren; Folaxin; FOLI-cell; Foliben; Folidan; Folidar; Folinac; Folinate Calcium; folinic acid; Folinic Acid Calcium Salt Pentahydrate; Folinoral; Folinvit; Foliplus; Folix; Imo; Lederfolat; Lederfolin; Leucosar; leucovorin; Rescufolin; Rescuvolin; Tonofolin; Wellcovorin
Drug: Mercaptopurine — Given PO
  Other Names: 3H-Purine-6-thiol; 6 MP; 6 Thiohypoxanthine; 6 Thiopurine; 6-Mercaptopurine; 6-Mercaptopurine Monohydrate; 6-MP; 6-Purinethiol; 6-Thiopurine; 6-Thioxopurine; 6H-Purine-6-thione, 1,7-dihydro- (9CI); 7-Mercapto-1,3,4,6-tetrazaindene; Alti-Mercaptopurine; Azathiopurine; Bw 57-323H; Flocofil; Ismipur; Leukerin; Leupurin; Mercaleukim; Mercaleukin; Mercaptina; Mercaptopurinum; Mercapurin; Mern; NCI-C04886; Puri-Nethol; Purimethol; Purine, 6-mercapto-; Purine-6-thiol (8CI); Purine-6-thiol, monohydrate; Purinethiol; Purinethol; U-4748; WR-2785
Drug: Methotrexate — Given IV, IT, or PO
  Other Names: Abitrexate; Alpha-Methopterin; Amethopterin; Brimexate; CL 14377; CL-14377; Emtexate; Emthexat; Emthexate; Farmitrexat; Fauldexato; Folex; Folex PFS; Lantarel; Ledertrexate; Lumexon; Maxtrex; Medsatrexate; Metex; Methoblastin; Methotrexate LPF; Methotrexate Methylaminopterin; Methotrexatum; Metotrexato; Metrotex; Mexate; Mexate-AQ; MTX; Novatrex; Rheumatrex; Texate; Tremetex; Trexeron; Trixilem; WR-19039
Drug: Methylprednisolone — Given IV
  Other Names: Adlone; Caberdelta M; DepMedalone; Depo Moderin; Depo-Nisolone; Duralone; Emmetipi; Esametone; Firmacort; Medlone 21; Medrate; Medrol; Medrol Veriderm; Medrone; Mega-Star; Meprolone; Methylprednisolonum; Metilbetasone Solubile; Metrocort; Metypresol; Metysolon; Predni-M-Tablinen; Prednilen; Radilem; Sieropresol; Solpredone; Summicort; Urbason; Veriderm Medrol; Wyacort
Procedure: Multigated Acquisition Scan — Undergo MUGA
  Other Names: Blood Pool Scan; Equilibrium Radionuclide Angiography; Gated Blood Pool Imaging; Gated Heart Pool Scan; MUGA; MUGA Scan; Multi-Gated Acquisition Scan; Radionuclide Ventriculogram Scan; Radionuclide Ventriculography; RNVG; SYMA Scanning; Synchronized Multigated Acquisition Scanning
Drug: Pegaspargase — Given IM
  Other Names: L-Asparaginase with Polyethylene Glycol; Oncaspar; Oncaspar-IV; PEG-Asparaginase; PEG-L-Asparaginase; PEG-L-Asparaginase (Enzon - Kyowa Hakko); PEGLA; Polyethylene Glycol L-Asparaginase; Polyethylene Glycol-L-Asparaginase
Other: Pharmacological Study — Correlative studies
Drug: Prednisone — Given PO
  Other Names: .delta.1-Cortisone; 1, 2-Dehydrocortisone; Adasone; Cortancyl; Dacortin; DeCortin; Decortisyl; Decorton; Delta 1-Cortisone; Delta-Dome; Deltacortene; Deltacortisone; Deltadehydrocortisone; Deltasone; Deltison; Deltra; Econosone; Lisacort; Meprosona-F; Metacortandracin; Meticorten; Ofisolona; Orasone; Panafcort; Panasol-S; Paracort; Perrigo Prednisone; PRED; Predicor; Predicorten; Prednicen-M; Prednicort; Prednidib; Prednilonga; Predniment; Prednisone Intensol; Prednisonum; Prednitone; Promifen; Rayos; Servisone; SK-Prednisone
Drug: Therapeutic Hydrocortisone — Given IT
  Other Names: Aeroseb-HC; Barseb HC; Barseb-HC; Cetacort; Cort-Dome; Cortef; Cortenema; Cortifan; Cortisol; Cortispray; Cortril; Dermacort; Domolene; Eldecort; Hautosone; Heb-Cort; Hydrocortisone; Hydrocortone; Hytone; Komed-HC; Nutracort; Proctocort; Rectoid
Drug: Vincristine Sulfate — Given IV
  Other Names: Kyocristine; Leurocristine Sulfate; Leurocristine, sulfate; Oncovin; Vincasar; Vincosid; Vincrex; Vincristine, sulfate

SUMMARY:
This phase III trial studies combination chemotherapy with or without lestaurtinib with to see how well they work in treating younger patients with newly diagnosed acute lymphoblastic leukemia. Drugs used in chemotherapy work in different ways to stop the growth of stop cancer cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Lestaurtinib may stop the growth of cancer cells by blocking some of the enzymes needed for cell growth. It is not yet known whether combination chemotherapy is more effective with or without lestaurtinib in treating acute lymphoblastic leukemia.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To estimate the 3-year event-free survival (EFS) of infants with mixed lineage leukemia-rearranged (MLL-R) acute lymphoblastic leukemia (ALL) treated with chemotherapy plus the fms-related tyrosine kinase 3 (FLT3) inhibitor lestaurtinib.

SECONDARY OBJECTIVES:

I. To compare the 3-year EFS of infants with MLL-R ALL treated with chemotherapy plus the FLT3 inhibitor lestaurtinib to MLL-R patients treated with chemotherapy alone.

II. To determine a safe, tolerable and biologically active dose of lestaurtinib given in sequential combination with chemotherapy in MLL-R infants.

III. To characterize the pharmacokinetics and pharmacodynamics of lestaurtinib in infants when given at the proposed dose in sequential combination with chemotherapy.

IV. To identify molecular mechanisms of resistance to lestaurtinib in leukemic blasts.

V. To describe levels of minimal residual disease in infants with ALL within the context of the proposed therapy, and correlate with outcome.

VI. To identify gene expression patterns in diagnostic infant leukemia samples that correlate with outcome within the context of the proposed therapy.

VII. To describe the outcome of infants with MLL-G ALL treated with a modified P9407 chemotherapy backbone that includes an extended continuation phase.

OUTLINE:

INDUCTION THERAPY (WEEKS 1-5): All patients receive induction therapy comprising vincristine sulfate intravenously (IV) over 1 minute on days 8, 15, 22, and 29; daunorubicin hydrochloride IV over 30 minutes on days 8 and 9; cyclophosphamide IV over 30 minutes every 12 hours on days 3 and 4 (closed as of 05/19/09); pegaspargase or asparaginase intramuscularly (IM) on days 15, 18, 22, 25, 29, and 33; prednisone orally (PO) thrice daily (TID) or methylprednisolone IV on days 1-7; dexamethasone IV or PO TID on days 8-28; cytarabine IV over 30 minutes on days 8-21; methotrexate intrathecally (IT) on days 1 and 29; cytarabine IT on day 15; hydrocortisone IT on days 15 and 29; and filgrastim IV or subcutaneously (SC) beginning on day 5 and continuing until blood counts recover. Standard-risk patients are non-randomly assigned to receive a less intensive chemotherapy regimen without lestaurtinib (post-induction therapy A). Patients undergo echocardiography (ECHO) or multigated acquisition scan (MUGA), blood sample collection and bone marrow biopsy on day 1 week 1.

POST-INDUCTION THERAPY A: (for standard-risk patients MLL-germline [G])

INDUCTION INTENSIFICATION (WEEKS 6-9): Patients receive high-dose methotrexate IV continuously over 24 hours on days 1 and 8; triple IT chemotherapy comprising methotrexate, cytarabine, and hydrocortisone on days 1 and 8; leucovorin calcium IV or PO every 6 hours beginning 42 hours after start of high-dose methotrexate and continuing until methotrexate level is < 0.1 uM; cyclophosphamide IV over 30 minutes on days 15-19; etoposide IV over 2 hours on days 15-19; and filgrastim IV or SC beginning on day 20 and continuing until blood counts recover. Patients in morphologic remission proceed to re-induction therapy. Patients may undergo bone marrow biopsy on day 1 week 6.

RE-INDUCTION (WEEKS 10-12): Patients receive vincristine sulfate IV over 1 minute on days 1, 8, and 15; daunorubicin hydrochloride IV over 30 minutes on days 1 and 2; cyclophosphamide IV over 30 minutes every 12 hours on days 3 and 4; pegaspargase or asparaginase IM on day 4; dexamethasone IV or PO twice daily (BID) on days 1-7 and 15-21; triple IT chemotherapy comprising methotrexate, cytarabine, and hydrocortisone on days 1 and 15; and filgrastim IV or SC beginning on day 5 and continuing until blood counts recover. Patients undergo ECHO or MUGA, blood sample collection and bone marrow biopsy on day 1 week 10.

CONSOLIDATION (WEEKS 13-19): Patients receive high-dose methotrexate IV continuously over 24 hours on days 1 and 8; leucovorin calcium IV every 6 hours beginning 42 hours after start of high-dose methotrexate and continuing until methotrexate level is < 0.1 uM; triple IT chemotherapy comprising methotrexate, cytarabine, and hydrocortisone on day 1; etoposide IV over 2 hours on days 15-19; cyclophosphamide IV over 30 minutes on days 15-19; high-dose cytarabine IV over 3 hours every 12 hours on days 29 and 30; pegaspargase or asparaginase IM on day 30; and filgrastim IV or SC beginning on day 20 and day 31 and continuing until blood counts recover.

CONTINUATION I (WEEKS 20-41): Patients receive vincristine sulfate IV on day 1 in weeks 20 and 24; dexamethasone IV or PO BID on days 1-5 in weeks 20, and 24; triple IT chemotherapy comprising methotrexate, cytarabine, and hydrocortisone on day 1 in weeks 20 and 24; methotrexate IV on day 1 in weeks 21-24 and 25-27; etoposide IV over 2 hours on day 1-5 in week 28; cyclophosphamide IV over 30 minutes on days 1-5 in week 28; mercaptopurine PO on days 1-7 in weeks 21-23 and 25-27; and filgrastim SC or IV beginning on day 6 in week 28 and continuing until blood counts recover. Patients may undergo bone marrow biopsy on day 1 week 20.

CONTINUATION II (WEEKS 42-104): Patients receive vincristine sulfate IV on days 1, 29, and 57; dexamethasone IV or PO BID on days 1-5, 29-33, and 57-61; methotrexate IT on day 1; methotrexate PO on days 8, 15, 22, 36, 43, 50, 64, 71, and 78; and mercaptopurine PO on days 8-28, 36-56, and 64-84. Treatment repeats every 12 weeks for 2 years from diagnosis.

A safety/activity phase is conducted separately for the intermediate-risk (IR) and high-risk (HR) patients to identify a safe, tolerable, and biologically active dose of lestaurtinib combined with chemotherapy backbone. Once a tolerable/active dose of lestaurtinib has been identified for IR patients, subsequent IR patients are eligible to proceed to an efficacy phase, where they are randomized (or non-randomly assigned as of 7/16/2014) to chemotherapy with or without lestaurtinib. HR patients separately proceed to the randomized efficacy phase if a tolerable/active dose is identified for the HR stratum. IR and HR patients are randomized (or non-randomly assigned as of 7/16/2014) to 1 of 2 post-induction therapy regimens (post-induction therapy B or C).

POST-INDUCTION THERAPY B: (chemotherapy only for IR/HR patients classified as MLL-R; age >= 90 days at diagnosis):

INDUCTION INTENSIFICATION (WEEKS 6-9): Patients receive high-dose methotrexate, leucovorin calcium, cyclophosphamide, etoposide, and filgrastim as in post-induction therapy A induction intensification. Patients in morphologic remission proceed to re-induction Patients undergo ECHO or MUGA, blood sample collection and bone marrow biopsy on day 1 week 6. (Retired as of 7/16/2014)

RE-INDUCTION (WEEKS 10-12): Patients receive vincristine sulfate, daunorubicin hydrochloride, cyclophosphamide, pegaspargase or asparaginase, dexamethasone, triple IT chemotherapy, and filgrastim as in post-induction therapy A re-induction. Patients undergo ECHO or MUGA, blood sample collection and bone marrow biopsy on day 1 week 10. (Retired as of 7/16/2014)

CONSOLIDATION (WEEKS 13-19): Patients receive high-dose methotrexate, leucovorin calcium, triple IT chemotherapy, etoposide, cyclophosphamide, high-dose cytarabine, pegaspargase or asparaginase, and filgrastim as in post-induction therapy A consolidation. (Retired as of 7/16/2014)

CONTINUATION I (WEEKS 20-49): Patients receive vincristine sulfate IV over 1 minute on day 1 in weeks 20, 24, 33, 37, and 46; dexamethasone PO or IV BID on days 1-5 in weeks 20, 24, 33, 37, and 46; triple IT chemotherapy on day 1 in weeks 20, 24, 33, 37, and 46; methotrexate IV on day 1 in weeks 21-23, 25-26 and 37-45; mercaptopurine PO on days 1-7 in weeks 21-23, 25-26 and 37-45; etoposide IV over 2 hours on days 1-5 in week 27; cyclophosphamide IV over 2 hours on days 1-5 in week 27: high-dose cytarabine IV over 3 hours every 12 hours on days 1 and 2 in week 30; pegaspargase or asparaginase IM on day 2 in week 30: and filgrastim SC or IV beginning on day 3 in weeks 30 and continuing until blood counts recover. Patients may undergo bone marrow biopsy on day 1 of weeks 20, 33 and 46. (Retired as of 7/16/2014)

CONTINUATION II (WEEKS 50-104): Patients receive vincristine sulfate, dexamethasone, IT methotrexate, methotrexate PO, and mercaptopurine PO as in post-induction therapy A continuation II. Treatment repeats every 12 weeks for 2 years from diagnosis. (Retired as of 7/16/2014)

POST-INDUCTION THERAPY C: (chemotherapy and lestaurtinib for IR/HR patients classified as MLL-R; age < 90 days at diagnosis)

INDUCTION INTENSIFICATION THERAPY (WEEKS 6-9): Patients receive high-dose methotrexate, leucovorin calcium, cyclophosphamide, etoposide, and filgrastim as in post-induction therapy B induction intensification. Patients also receive lestaurtinib PO BID on days 20-27. Patients in morphologic remission proceed to re-induction.Patients undergo ECHO or MUGA, blood sample collection and bone marrow biopsy on day 1 week 6.

RE-INDUCTION (WEEKS 10-12): Patients receive vincristine sulfate, daunorubicin hydrochloride, cyclophosphamide, pegaspargase or asparaginase, dexamethasone, triple IT chemotherapy, and filgrastim as in post-induction therapy B re-induction. Patients also receive lestaurtinib PO on days 5-20. Patients undergo ECHO or MUGA, blood sample collection and bone marrow biopsy on day 1 week 10.

CONSOLIDATION (WEEKS 13-19) Patients receive high-dose methotrexate, leucovorin calcium, triple IT chemotherapy, etoposide, cyclophosphamide, high-dose cytarabine, pegaspargase or asparaginase, and filgrastim as in post-induction therapy B consolidation. Patients also receive lestaurtinib PO on days 20-27 and 31-42.

CONTINUATION I (WEEKS 20-49): Patients receive vincristine sulfate, dexamethasone, triple IT chemotherapy, methotrexate, mercaptopurine, etoposide, high-dose cytarabine, pegaspargase or asparaginase, and filgrastim as in post-induction therapy B continuation I. Patients also receive lestaurtinib PO on days 2-6 in weeks 20 and 24; days 27-41 in weeks 27-29; days 45-56 in weeks 30-32. Patients may undergo bone marrow biopsy on day 1 of weeks 20, 33 and 46.

CONTINUATION II (WEEKS 50-104): Patients receive vincristine sulfate, dexamethasone, IT methotrexate, methotrexate PO, and mercaptopurine PO as in post-induction therapy B continuation II. Treatment repeats every 12 weeks for 2 years from diagnosis.

After completion of study treatment, all patients are followed up every 1-6 months for 4 years and then annually thereafter.

ELIGIBILITY:
Inclusion Criteria:

* Patients must be enrolled on a Children's Oncology Group (COG) ALL Classification Study (AALL08B1) prior to enrollment on AALL0631
* Patients must be < 366 days of age at the time of diagnosis; for neonates in the first month of life, patients must be > 36 weeks gestational age at the time of diagnosis
* Patients must be newly diagnosed with acute lymphoblastic leukemia (ALL) or acute undifferentiated leukemia (AUL); patients with T-cell ALL are eligible; patients with bilineage or biphenotypic acute leukemia are eligible, provided the morphology and immunophenotype are predominately lymphoid
* Patients must be previously untreated with the exception of steroids and intrathecal chemotherapy; no other systemic chemotherapy may have been administered; patients receiving prior steroid therapy are eligible for study; any amount of steroid pretreatment will not affect initial induction assignment as long as the patient meets all other eligibility criteria; IT chemotherapy per protocol is allowed for patient convenience at the time of the diagnostic bone marrow or venous line placement to avoid second lumbar puncture; (note: the central nervous system [CNS] status must be determined based on a sample obtained prior to administration of any systemic or intrathecal chemotherapy, except for steroid pretreatment); systemic chemotherapy must begin within 72 hours of this IT therapy
* All patients and/or their parents or legal guardians must sign a written informed consent
* All institutional, Food and Drug Administration (FDA), and National Cancer Institute (NCI) requirements for human studies must be met
* Patients with mature B-cell ALL or acute myelogenous leukemia (AML) are NOT eligible
* Patients with Down syndrome are NOT eligible

Max Age: 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 218 (Actual)
Dates: Start 2008-01-15 (Actual); Primary Completion 2017-09-30 (Actual); Study Completion 2024-06-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joanne M Hilden, Principal Investigator — Children's Oncology Group
Locations (170):
- United States (157):
  - Children's Hospital of Alabama, Birmingham, Alabama
  - University of Alabama at Birmingham Cancer Center, Birmingham, Alabama
  - Phoenix Childrens Hospital, Phoenix, Arizona
  - Arkansas Children's Hospital, Little Rock, Arkansas
  - University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - Kaiser Permanente Downey Medical Center, Downey, California
  - Loma Linda University Medical Center, Loma Linda, California
  - Miller Children's and Women's Hospital Long Beach, Long Beach, California
  - Cedars Sinai Medical Center, Los Angeles, California
  - Valley Children's Hospital, Madera, California
  - UCSF Benioff Children's Hospital Oakland, Oakland, California
  - Kaiser Permanente-Oakland, Oakland, California
  - Children's Hospital of Orange County, Orange, California
  - Lucile Packard Children's Hospital Stanford University, Palo Alto, California
  - University of California Davis Comprehensive Cancer Center, Sacramento, California
  - Rady Children's Hospital - San Diego, San Diego, California
  - UCSF Medical Center-Parnassus, San Francisco, California
  - UCSF Medical Center-Mission Bay, San Francisco, California
  - Children's Hospital Colorado, Aurora, Colorado
  - Rocky Mountain Hospital for Children-Presbyterian Saint Luke's Medical Center, Denver, Colorado
  - Connecticut Children's Medical Center, Hartford, Connecticut
  - Yale University, New Haven, Connecticut
  - Alfred I duPont Hospital for Children, Wilmington, Delaware
  - MedStar Georgetown University Hospital, Washington D.C., District of Columbia
  - Children's National Medical Center, Washington D.C., District of Columbia
  - Lee Memorial Health System, Fort Myers, Florida
  - Golisano Children's Hospital of Southwest Florida, Fort Myers, Florida
  - University of Florida Health Science Center - Gainesville, Gainesville, Florida
  - Nemours Children's Clinic-Jacksonville, Jacksonville, Florida
  - University of Miami Miller School of Medicine-Sylvester Cancer Center, Miami, Florida
  - Miami Cancer Institute, Miami, Florida
  - AdventHealth Orlando, Orlando, Florida
  - Arnold Palmer Hospital for Children, Orlando, Florida
  - Nemours Children's Clinic - Orlando, Orlando, Florida
  - Orlando Health Cancer Institute, Orlando, Florida
  - Nemours Children's Hospital, Orlando, Florida
  - Nemours Children's Clinic - Pensacola, Pensacola, Florida
  - Johns Hopkins All Children's Hospital, St. Petersburg, Florida
  - Saint Joseph's Hospital/Children's Hospital-Tampa, Tampa, Florida
  - Saint Mary's Hospital, West Palm Beach, Florida
  - Children's Healthcare of Atlanta - Egleston, Atlanta, Georgia
  - Augusta University Medical Center, Augusta, Georgia
  - Memorial Health University Medical Center, Savannah, Georgia
  - University of Hawaii Cancer Center, Honolulu, Hawaii
  - Kapiolani Medical Center for Women and Children, Honolulu, Hawaii
  - Tripler Army Medical Center, Honolulu, Hawaii
  - Saint Luke's Cancer Institute - Boise, Boise, Idaho
  - Lurie Children's Hospital-Chicago, Chicago, Illinois
  - University of Illinois, Chicago, Illinois
  - University of Chicago Comprehensive Cancer Center, Chicago, Illinois
  - Loyola University Medical Center, Maywood, Illinois
  - Advocate Children's Hospital-Oak Lawn, Oak Lawn, Illinois
  - Advocate Children's Hospital-Park Ridge, Park Ridge, Illinois
  - Advocate Lutheran General Hospital, Park Ridge, Illinois
  - Riley Hospital for Children, Indianapolis, Indiana
  - Ascension Saint Vincent Indianapolis Hospital, Indianapolis, Indiana
  - Blank Children's Hospital, Des Moines, Iowa
  - University of Kentucky/Markey Cancer Center, Lexington, Kentucky
  - Norton Children's Hospital, Louisville, Kentucky
  - Tulane University School of Medicine, New Orleans, Louisiana
  - Children's Hospital New Orleans, New Orleans, Louisiana
  - Eastern Maine Medical Center, Bangor, Maine
  - University of Maryland/Greenebaum Cancer Center, Baltimore, Maryland
  - Sinai Hospital of Baltimore, Baltimore, Maryland
  - Johns Hopkins University/Sidney Kimmel Cancer Center, Baltimore, Maryland
  - Tufts Children's Hospital, Boston, Massachusetts
  - C S Mott Children's Hospital, Ann Arbor, Michigan
  - Wayne State University/Karmanos Cancer Institute, Detroit, Michigan
  - Michigan State University Clinical Center, East Lansing, Michigan
  - Hurley Medical Center, Flint, Michigan
  - Corewell Health Grand Rapids Hospitals - Helen DeVos Children's Hospital, Grand Rapids, Michigan
  - Bronson Methodist Hospital, Kalamazoo, Michigan
  - Kalamazoo Center for Medical Studies, Kalamazoo, Michigan
  - Children's Hospitals and Clinics of Minnesota - Minneapolis, Minneapolis, Minnesota
  - University of Minnesota/Masonic Cancer Center, Minneapolis, Minnesota
  - Mayo Clinic in Rochester, Rochester, Minnesota
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Columbia Regional, Columbia, Missouri
  - Children's Mercy Hospitals and Clinics, Kansas City, Missouri
  - Mercy Hospital Saint Louis, St Louis, Missouri
  - Children's Hospital and Medical Center of Omaha, Omaha, Nebraska
  - Alliance for Childhood Diseases/Cure 4 the Kids Foundation, Las Vegas, Nevada
  - Summerlin Hospital Medical Center, Las Vegas, Nevada
  - Nevada Cancer Research Foundation NCORP, Las Vegas, Nevada
  - Dartmouth Hitchcock Medical Center/Dartmouth Cancer Center, Lebanon, New Hampshire
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Saint Barnabas Medical Center, Livingston, New Jersey
  - Morristown Medical Center, Morristown, New Jersey
  - Saint Peter's University Hospital, New Brunswick, New Jersey
  - Rutgers Cancer Institute of New Jersey-Robert Wood Johnson University Hospital, New Brunswick, New Jersey
  - Newark Beth Israel Medical Center, Newark, New Jersey
  - Saint Joseph's Regional Medical Center, Paterson, New Jersey
  - Overlook Hospital, Summit, New Jersey
  - University of New Mexico Cancer Center, Albuquerque, New Mexico
  - Albany Medical Center, Albany, New York
  - Roswell Park Cancer Institute, Buffalo, New York
  - NYU Langone Hospital - Long Island, Mineola, New York
  - The Steven and Alexandra Cohen Children's Medical Center of New York, New Hyde Park, New York
  - Laura and Isaac Perlmutter Cancer Center at NYU Langone, New York, New York
  - University of Rochester, Rochester, New York
  - State University of New York Upstate Medical University, Syracuse, New York
  - Montefiore Medical Center - Moses Campus, The Bronx, New York
  - New York Medical College, Valhalla, New York
  - Mission Hospital, Asheville, North Carolina
  - UNC Lineberger Comprehensive Cancer Center, Chapel Hill, North Carolina
  - Carolinas Medical Center/Levine Cancer Institute, Charlotte, North Carolina
  - Novant Health Presbyterian Medical Center, Charlotte, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - East Carolina University, Greenville, North Carolina
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - Sanford Broadway Medical Center, Fargo, North Dakota
  - Children's Hospital Medical Center of Akron, Akron, Ohio
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Rainbow Babies and Childrens Hospital, Cleveland, Ohio
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Nationwide Children's Hospital, Columbus, Ohio
  - Dayton Children's Hospital, Dayton, Ohio
  - ProMedica Toledo Hospital/Russell J Ebeid Children's Hospital, Toledo, Ohio
  - Mercy Children's Hospital, Toledo, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Legacy Emanuel Children's Hospital, Portland, Oregon
  - Legacy Emanuel Hospital and Health Center, Portland, Oregon
  - Geisinger Medical Center, Danville, Pennsylvania
  - Penn State Children's Hospital, Hershey, Pennsylvania
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Saint Christopher's Hospital for Children, Philadelphia, Pennsylvania
  - Children's Hospital of Pittsburgh of UPMC, Pittsburgh, Pennsylvania
  - Rhode Island Hospital, Providence, Rhode Island
  - Prisma Health Richland Hospital, Columbia, South Carolina
  - BI-LO Charities Children's Cancer Center, Greenville, South Carolina
  - Greenville Cancer Treatment Center, Greenville, South Carolina
  - Sanford USD Medical Center - Sioux Falls, Sioux Falls, South Dakota
  - East Tennessee Childrens Hospital, Knoxville, Tennessee
  - Vanderbilt University/Ingram Cancer Center, Nashville, Tennessee
  - Texas Tech University Health Sciences Center-Amarillo, Amarillo, Texas
  - Dell Children's Medical Center of Central Texas, Austin, Texas
  - Driscoll Children's Hospital, Corpus Christi, Texas
  - Medical City Dallas Hospital, Dallas, Texas
  - UT Southwestern/Simmons Cancer Center-Dallas, Dallas, Texas
  - Cook Children's Medical Center, Fort Worth, Texas
  - Baylor College of Medicine/Dan L Duncan Comprehensive Cancer Center, Houston, Texas
  - Covenant Children's Hospital, Lubbock, Texas
  - Methodist Children's Hospital of South Texas, San Antonio, Texas
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas
  - Scott and White Memorial Hospital, Temple, Texas
  - Primary Children's Hospital, Salt Lake City, Utah
  - University of Vermont and State Agricultural College, Burlington, Vermont
  - Inova Fairfax Hospital, Falls Church, Virginia
  - Children's Hospital of The King's Daughters, Norfolk, Virginia
  - Providence Sacred Heart Medical Center and Children's Hospital, Spokane, Washington
  - Mary Bridge Children's Hospital and Health Center, Tacoma, Washington
  - Madigan Army Medical Center, Tacoma, Washington
  - West Virginia University Charleston Division, Charleston, West Virginia
  - Saint Vincent Hospital Cancer Center Green Bay, Green Bay, Wisconsin
  - University of Wisconsin Carbone Cancer Center - University Hospital, Madison, Wisconsin
  - Marshfield Medical Center-Marshfield, Marshfield, Wisconsin
  - Children's Hospital of Wisconsin, Milwaukee, Wisconsin
- Princess Margaret Hospital for Children, Perth, Western Australia, Australia
- Canada (11):
  - Alberta Children's Hospital, Calgary, Alberta
  - University of Alberta Hospital, Edmonton, Alberta
  - British Columbia Children's Hospital, Vancouver, British Columbia
  - CancerCare Manitoba, Winnipeg, Manitoba
  - Janeway Child Health Centre, St. John's, Newfoundland and Labrador
  - IWK Health Centre, Halifax, Nova Scotia
  - Children's Hospital, London, Ontario
  - Children's Hospital of Eastern Ontario, Ottawa, Ontario
  - Hospital for Sick Children, Toronto, Ontario
  - The Montreal Children's Hospital of the MUHC, Montreal, Quebec
  - Saskatoon Cancer Centre, Saskatoon, Saskatchewan
- Starship Children's Hospital, Grafton, Auckland, New Zealand

IPD SHARING:
Plan to Share IPD: Yes
Select individual patient-level data from this trial can be requested from the NCTN/NCORP Data Archive

REFERENCES:
- [Derived] Loftus JP, Yahiaoui A, Brown PA, Niswander LM, Bagashev A, Wang M, Schauf A, Tannheimer S, Tasian SK. Combinatorial efficacy of entospletinib and chemotherapy in patient-derived xenograft models of infant acute lymphoblastic leukemia. Haematologica. 2021 Apr 1;106(4):1067-1078. doi: 10.3324/haematol.2019.241729. PMID 32414848
- See also: Data Available: Select individual patient-level data from this trial can be requested from the NCTN/NCORP Data Archive — https://nctn-data-archive.nci.nih.gov/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Infants with Acute Lymphoblastic Leukemia (ALL)
Pre-assignment Details: MLL-germline [G] to SR (Arm A/Group 1), MLL-rearranged [R] randomized/assigned to Arm B (Group2; chemo) or Arm C (Group3; chemo+lestaurtinib) with dose determined by age at dx (>=90 days is IR and <90 days is HR)
Groups:
- Induction (All Patients): All Patients for Induction (not assigned).
- Arm A (Standard Risk MLL-G): Eligible patients with MLL-G (germline, or non-rearranged)
  Asparaginase: Given IV, IM, or PO
  Cyclophosphamide: Given IV
  Cytarabine: Given IV or IT
  Daunorubicin Hydrochloride: Given IV
  Dexamethasone: Given IV or PO
  Etoposide: Given IV
  Filgrastim: Given IV or SC
  Laboratory Biomarker Analysis: Correlative studies
  Leucovorin Calcium: Given IV
  Mercaptopurine: Given PO
  Methotrexate: Given IV, IT, or PO
  Methylprednisolone: Given IV
  Pegaspargase: Given IM
  Pharmacological Study: Correlative studies
  Prednisone: Given PO
  Therapeutic Hydrocortisone: Given IT
  Vincristine Sulfate: Given IV
- Arm B (IR/HR MLL-R Chemotherapy): Eligible patients with MLL-R (rearranged). Considered Intermediate Risk (IR) if age >= 90 days at diagnosis and High Risk (HR) if age < 90 days at diagnosis.
  Asparaginase: Given IV, IM, or PO
  Cyclophosphamide: Given IV
  Cytarabine: Given IV or IT
  Daunorubicin Hydrochloride: Given IV
  Dexamethasone: Given IV or PO
  Etoposide: Given IV
  Filgrastim: Given IV or SC
  Laboratory Biomarker Analysis: Correlative studies
  Leucovorin Calcium: Given IV
  Mercaptopurine: Given PO
  Methotrexate: Given IV, IT, or PO
  Methylprednisolone: Given IV
  Pegaspargase: Given IM
  Pharmacological Study: Correlative studies
  Prednisone: Given PO
  Therapeutic Hydrocortisone: Given IT
  Vincristine Sulfate: Given IV
- Arm C (Safety/ Dose Level 1): Arm C, IR/HR MLL-R chemotherapy and lestaurtinib at Dose Level 1 (DL1) (HR: 3.5 mg/kg/day; SR: 4 mg/kg/day)
- ARM C (Safety/ Dose Level 2): Arm C, IR/HR MLL-R chemotherapy and lestaurtinib at Dose Level 2 (DL2) (HR: 4.25 mg/kg/day; SR: 5 mg/kg/day)
- Arm C (Efficacy/ Dose Level 2): Arm C, IR/HR MLL-R chemotherapy and lestaurtinib at Dose Level 2 (DL2)-Efficacy (HR: 4.25 mg/kg/day; SR: 5 mg/kg/day)
Period: Induction
Arm/Group | Induction (All Patients) | Arm A (Standard Risk MLL-G) | Arm B (IR/HR MLL-R Chemotherapy) | Arm C (Safety/ Dose Level 1) | ARM C (Safety/ Dose Level 2) | Arm C (Efficacy/ Dose Level 2)
Started | 218 | 0 | 0 | 0 | 0 | 0
Completed | 192 | 0 | 0 | 0 | 0 | 0
Not Completed | 26 | 0 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 2 | 0 | 0 | 0 | 0 | 0
Not completed — Death | 6 | 0 | 0 | 0 | 0 | 0
Not completed — Physician Decision | 3 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Refusal of Further Protocol Therapy | 2 | 0 | 0 | 0 | 0 | 0
Not completed — Ineligible | 8 | 0 | 0 | 0 | 0 | 0
Not completed — Inevaluable for post Induction | 2 | 0 | 0 | 0 | 0 | 0
Not completed — Unable to receive Lestaurtinib-Not in US | 2 | 0 | 0 | 0 | 0 | 0
Period: Post Induction Therapy by Tx Assignment
Arm/Group | Induction (All Patients) | Arm A (Standard Risk MLL-G) | Arm B (IR/HR MLL-R Chemotherapy) | Arm C (Safety/ Dose Level 1) | ARM C (Safety/ Dose Level 2) | Arm C (Efficacy/ Dose Level 2)
Started | 0 | 60 | 54 | 11 | 11 | 56
Completed | 0 | 50 | 22 | 4 | 4 | 19
Not Completed | 0 | 10 | 32 | 7 | 7 | 37
Not completed — Adverse Event | 0 | 1 | 2 | 1 | 0 | 3
Not completed — Death | 0 | 0 | 2 | 0 | 2 | 2
Not completed — Physician Decision | 0 | 3 | 5 | 1 | 2 | 2
Not completed — Refusal of Further Protocol | 0 | 1 | 0 | 2 | 2 | 5
Not completed — Relapse | 0 | 5 | 16 | 3 | 1 | 20
Not completed — Developed second malignant neoplasm | 0 | 0 | 1 | 0 | 0 | 0
Not completed — Patient Moved to Another Institution | 0 | 0 | 2 | 0 | 0 | 0
Not completed — Induction Failure | 0 | 0 | 4 | 0 | 0 | 5

BASELINE CHARACTERISTICS:
Groups:
- All Patients: All patients for Induction
Arm/Group | All Patients
Number analyzed (Participants) | 218
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 218
  Between 18 and 65 years | 0
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: Years] | 0.54 (0.28)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 122
  Male | 96
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 50
  Not Hispanic or Latino | 160
  Unknown or Not Reported | 8
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 3
  Asian | 9
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 16
  White | 167
  More than one race | 0
  Unknown or Not Reported | 23
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 201
  Canada | 15
  New Zealand | 1
  Australia | 1

OUTCOME MEASURES:

1. Primary Outcome: Percent Probability for Event-free Survival (EFS) for Patients on Arm C at Dose Level 2 (DL2)
Description: EFS time is defined as time from randomization to first event (relapse, second malignant neoplasm, death) or date of last contact for patients who are event-free. EFS is constructed using the Kaplan-Meier life table method with confidence interval based on standard errors computed using the method of Peto and Peto.
Time Frame: From start of post-induction therapy for up to 10 years
Population: All 67 patients on Arm C (Safety and Efficacy at Dose Level 2) were included in the analysis.
Measure: Number (90% Confidence Interval); unit: percentage probability
Groups:
- Arm C (Safety/Efficacy Dose Level 2): Arm C (Safety and Efficacy), IR/HR MLL-R chemotherapy and lestaurtinib at DL2 (HR: 4.25 mg/kg/day; SR: 5 mg/kg/day)
Arm/Group | Arm C (Safety/Efficacy Dose Level 2)
Number analyzed (Participants) | 67
percentage probability | 35.82 [25.98 to 45.66]

2. Secondary Outcome: Percent Probability for Event-free Survival (EFS) of MLL-R Infants Treated With Combination Chemotherapy With or Without Lestaurtinib at DL2
Description: Event Free Probability where EFS time is defined as time from randomization to first event (relapse, second malignant neoplasm, death) or date of last contact for patients who are event-free. EFS is constructed using the Kaplan-Meier life table method with confidence interval based on standard errors computed using the method of Peto and Peto. EFS will be compared between patients on treatment Arm C at DL2 to those on Arm B.
Time Frame: From start of post-induction therapy for up to 10 years.
Population: All eligible Arm B and ARM C (Dose Level 2) patients were included in the analysis.
Measure: Number (90% Confidence Interval); unit: percent probability
Groups:
- Arm C (IR/HR MLL-R Chemotherapy and Lestaurtinib): Eligible patients with MLL-R (rearranged). Considered Intermediate Risk (IR) if age >= 90 days at diagnosis and High Risk (HR) if age < 90 days at diagnosis.
  Asparaginase: Given IV, IM, or PO
  Cyclophosphamide: Given IV
  Cytarabine: Given IV or IT
  Daunorubicin Hydrochloride: Given IV
  Dexamethasone: Given IV or PO
  Etoposide: Given IV
  Filgrastim: Given IV or SC
  Laboratory Biomarker Analysis: Correlative studies
  Lestaurtinib: Given PO
  Leucovorin Calcium: Given IV
  Mercaptopurine: Given PO
  Methotrexate: Given IV, IT, or PO
  Methylprednisolone: Given IV
  Pegaspargase: Given IM
  Pharmacological Study: Correlative studies
  Prednisone: Given PO
  Therapeutic Hydrocortisone: Given IT
  Vincristine Sulfate: Given IV
Arm/Group | Arm B (IR/HR MLL-R Chemotherapy) | Arm C (IR/HR MLL-R Chemotherapy and Lestaurtinib)
Number analyzed (Participants) | 54 | 67
percent probability | 38.89 [27.98 to 49.80] | 35.82 [25.98 to 45.66]
Statistical Analysis 1: Comparison: Arm B (IR/HR MLL-R Chemotherapy) vs Arm C (IR/HR MLL-R Chemotherapy and Lestaurtinib); A one-sided log rank test will be used for testing whether the EFS in Arm C (chemo+lest) at DL2 is greater than the EFS in Arm B (chemo). This is equivalent to testing the null hypothesis of hazard ratio (HR)=1 versus the alternative of HR<1; Test type: Superiority; p = 0.672, Log Rank — A priori significance level threshold of alpha=0.15; Hazard Ratio (HR) = 1.107, 85% CI 1-sided [upper limit 1.403] — Arm C is the numerator and Arm B is the denominator of the estimated hazard ratio

3. Secondary Outcome: Number of Patients Who Experienced Lestaurtinib-related Dose Limiting Toxicity (DLT)
Description: Lestaurtinib-related dose-limiting toxicity proportions, as measured by NCI Common Terminology Criteria for Adverse Events (CTCAE) version 4.0, will by summarized by dose level for Safety phase patients.
Time Frame: Up to 12 weeks from start of induction
Population: Arm C patients of Safety Phase who were evaluable for DLT. The first 10 evaluable patients enrolled on each dose level were included for monitoring dose limiting toxicity.
Measure: Count of Participants; unit: Participants
Groups:
- Arm C (IR/HR MLL-R Chemotherapy and Lestaurtinib-Dose Level 1): Evaluable Arm C, IR/HR MLL-R chemotherapy and lestaurtinib at DL1 (HR: 3.5 mg/kg/day; SR: 4 mg/kg/day)
- Arm C (IR/HR MLL-R Chemotherapy and Lestaurtinib-Dose Level 2): Evaluable Arm C, IR/HR MLL-R chemotherapy and lestaurtinib at DL2 (HR: 4.25 mg/kg/day; SR: 5 mg/kg/day)
Arm/Group | Arm C (IR/HR MLL-R Chemotherapy and Lestaurtinib-Dose Level 1) | Arm C (IR/HR MLL-R Chemotherapy and Lestaurtinib-Dose Level 2)
Number analyzed (Participants) | 10 | 10
Participants | 0 | 1

4. Secondary Outcome: Pharmacokinetic AGP Levels in Infants Given Lestaurtinib at DL2 in Combination With Chemotherapy
Description: Pharmacokinetic AGP levels in infants given lestaurtinib at DL2 in combination with chemotherapy will be described with mean and standard deviation for those with available data.
Time Frame: Up to 12 weeks
Population: Data was and never will be collected
Arm/Group | Arm C (IR/HR MLL-R Chemotherapy and Lestaurtinib)
Number analyzed (Participants) | 0

5. Secondary Outcome: Pharmacokinetic Albumin in Infants Given Lestaurtinib at DL2 in Combination With Chemotherapy
Description: Pharmacokinetic albumin in infants given lestaurtinib at DL2 in combination with chemotherapy will be described with mean and standard deviation for those with available data.
Time Frame: Up to 12 weeks
Population: Data was and never will be collected
Arm/Group | Arm C (IR/HR MLL-R Chemotherapy and Lestaurtinib)
Number analyzed (Participants) | 0

6. Secondary Outcome: Pharmacodynamics PIA Levels in Infants Given Lestaurtinib at DL2 in Combination With Chemotherapy
Description: Summarized with mean and standard deviation for those with available data in Arm C
Time Frame: Sampled between weeks 6-12 from start of induction
Population: Arm C Dose Level 2 (DL2) patients who had data available for analysis.
Measure: Mean (Standard Deviation); unit: Activity percentage
Arm/Group | Arm C (Safety/Efficacy Dose Level 2)
Number analyzed (Participants) | 63
Activity percentage | 69.00 (22.96)

7. Secondary Outcome: Describe FLT3 Protein Expression as a Molecular Mechanism of Primary Resistance to Lestaurtinib in Leukemic Blasts
Description: Described via mean and standard deviation by group.
Time Frame: Sampled at the start of induction
Population: Patients who had data collected
Measure: Mean (Standard Deviation); unit: qPCR fold expression ratio
Arm/Group | Arm A (Standard Risk MLL-G) | Arm B (IR/HR MLL-R Chemotherapy) | Arm C (IR/HR MLL-R Chemotherapy and Lestaurtinib)
Number analyzed (Participants) | 51 | 38 | 65
qPCR fold expression ratio | 1.25 (2.12) | 7.85 (10.65) | 5.83 (5.55)

8. Secondary Outcome: Describe FLT3 Protein Expression as a Molecular Mechanism of Acquired Resistance to Lestaurtinib in Leukemic Blasts
Description: Described via means and standard deviations in available Arm C relapse samples
Time Frame: At relapse (up to 3 years)
Population: Arm C Dose Level 2 patients who relapsed and had data collected.
Measure: Mean (Standard Deviation); unit: qPCR fold expression ratio
Arm/Group | Arm C (Safety/Efficacy Dose Level 2)
Number analyzed (Participants) | 7
qPCR fold expression ratio | 5.73 (4.56)

9. Secondary Outcome: Describe in Vitro Sensitivity as a Molecular Mechanism of Primary Resistance to Lestaurtinib in Leukemic Blasts
Description: Described via means and standard deviations in samples which have primary resistance to lestaurtinib
Time Frame: Sampled at the start of induction
Population: Patients who had data collected
Measure: Median (Standard Deviation); unit: Proportion of cells that are viable
Arm/Group | Arm A (Standard Risk MLL-G) | Arm B (IR/HR MLL-R Chemotherapy) | Arm C (IR/HR MLL-R Chemotherapy and Lestaurtinib)
Number analyzed (Participants) | 43 | 37 | 62
Proportion of cells that are viable | 0.75 (0.14) | 0.48 (0.19) | 0.47 (0.19)

10. Secondary Outcome: Describe in Vitro Sensitivity as a Molecular Mechanism of Acquired Resistance to Lestaurtinib in Leukemic Blasts
Description: Described via means and standard deviations in samples which have acquired resistance to lestaurtinib
Time Frame: At relapse (up to 3 years)
Population: Arm C Dose Level 2 patients who relapsed and had data collected
Measure: Mean (Standard Deviation); unit: Proportion of cells that are viable
Arm/Group | Arm C (IR/HR MLL-R Chemotherapy and Lestaurtinib)
Number analyzed (Participants) | 7
Proportion of cells that are viable | 0.69 (0.15)

11. Secondary Outcome: Percent Probability of Event Free Survival (EFS) by MRD Status and Treatment Arm
Description: Three-year EFS estimates and 90% CI will be reported by treatment arm and end-induction MRD status.
Time Frame: 3 Years from end of Induction)
Population: Patients who had data collected
Measure: Number (90% Confidence Interval); unit: percent probability
Groups:
- Arm A (MRD Negative); Arm A (MRD Positive): Arm A, standard risk MLL-G
- Arm B (MRD Negative); Arm B (MRD Positive): Arm B, IR/HR MLL-R chemotherapy
- Arm C (MRD Negative); Arm C (MRD Positive): Arm C, IR/HR MLL-R chemotherapy and lestaurtinib
Arm/Group | Arm A (MRD Negative) | Arm A (MRD Positive) | Arm B (MRD Negative) | Arm B (MRD Positive) | Arm C (MRD Negative) | Arm C (MRD Positive)
Number analyzed (Participants) | 43 | 8 | 19 | 22 | 27 | 37
percent probability | 86.05 [77.36 to 94.74] | 87.5 [68.27 to 100] | 47.37 [28.53 to 66.21] | 22.73 [8.04 to 37.42] | 51.85 [36.03 to 67.67] | 27.03 [13.61 to 40.45]

12. Secondary Outcome: Identification of Gene Expression Patterns in Diagnostic Infant Leukemia Samples That Correlate With Survival Outcomes
Description: EFS outcomes will be reported by genotype.
Time Frame: At 3 years
Population: Data was and never will never be collected.
Arm/Group | Arm A (Standard Risk MLL-G) | Arm B (IR/HR MLL-R Chemotherapy) | Arm C (IR/HR MLL-R Chemotherapy and Lestaurtinib)
Number analyzed (Participants) | 0 | 0 | 0

13. Secondary Outcome: Identification of Gene Expression Patterns in Diagnostic Infant Leukemia Samples That Correlate With PIA Values
Description: Means and standard deviations of Plasma Inhibitory Activity (PIA) will be given by genotype
Time Frame: At 3 years
Population: Data was and never will be collected
Arm/Group | Arm A (Standard Risk MLL-G) | Arm B (IR/HR MLL-R Chemotherapy) | Arm C (IR/HR MLL-R Chemotherapy and Lestaurtinib)
Number analyzed (Participants) | 0 | 0 | 0

14. Secondary Outcome: Percent Probability for Event-free Survival (EFS) for Patients on Arm A
Description: EFS time is defined as time from treatment assignment to first event (relapse, second malignant neoplasm, death) or date of last contact for patients who are event-free. EFS is constructed using the Kaplan-Meier life table method with confidence interval based on standard errors computed using the method of Peto and Peto.
Time Frame: From start of post-induction therapy for up to 10 years
Population: All Eligible patients treated in Arm A (standard risk MLL-G).
Measure: Number (90% Confidence Interval); unit: percentage probability
Arm/Group | Arm A (Standard Risk MLL-G)
Number analyzed (Participants) | 60
percentage probability | 86.67 [79.45 to 93.89]

ADVERSE EVENTS:
Time Frame: Group 1: Study Entry to end-Induction (5 weeks). Other Groups: Start of Induction Intensification (Week 6) through 10 years post study enrollment.
Description: Adverse event reporting is collected routinely using case report forms. SAE field contains NCI Common Terminology Criteria for Adverse Events (CTCAEs) submitted via expedited reporting (NCI AdEERs / CAeRs). The AE field contains grade 3 and higher CTCAEs reported on study excluding those that were reported as SAEs. Ineligible patients are excluded from reporting of adverse events.
Groups:
- Post Induction (Follow-up Only): Post-Induction patients that did not receive therapy
Arm/Group | Induction (All Patients) | Post Induction (Follow-up Only) | Arm A (Standard Risk MLL-G) | Arm B (IR/HR MLL-R Chemotherapy) | Arm C (Safety/ Dose Level 1) | Arm C (Safety/ Dose Level 2) | Arm C (Efficacy/ Dose Level 2)
All-Cause Mortality (participants affected / at risk) | 6/210 | 6/12 | 3/60 | 31/54 | 6/11 | 5/11 | 28/56
Serious Adverse Events (participants affected / at risk) | 9/210 | 0/12 | 2/60 | 9/54 | 8/11 | 7/11 | 41/56
Other Adverse Events (participants affected / at risk) | 181/210 | 5/12 | 59/60 | 54/54 | 11/11 | 11/11 | 55/56
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Induction (All Patients) (N=210) | Post Induction (Follow-up Only) (N=12) | Arm A (Standard Risk MLL-G) (N=60) | Arm B (IR/HR MLL-R Chemotherapy) (N=54) | Arm C (Safety/ Dose Level 1) (N=11) | Arm C (Safety/ Dose Level 2) (N=11) | Arm C (Efficacy/ Dose Level 2) (N=56)
Anemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 2 (5)
Blood and lymphatic system disorders - Other, specify (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 6 (7) | 1 (1) | 22 (42)
Hemolytic uremic syndrome (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Thrombotic thrombocytopenic purpura (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cardiac arrest (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Heart failure (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Left ventricular systolic dysfunction (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Myocarditis (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3)
Ascites (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Colitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 3 (6)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 5 (9) | 3 (3) | 11 (14)
Enterocolitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Gastric hemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gastrointestinal disorders - Other, specify (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 5 (5)
Gastrointestinal fistula (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Lower gastrointestinal hemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Mucositis oral (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 2 (3) | 9 (11)
Oral pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Small intestinal perforation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Typhlitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Death NOS (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Fatigue (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Fever (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 3 (4)
General disorders and administration site conditions - Other, specify (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Irritability (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Multi-organ failure (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Anaphylaxis (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Immune system disorders - Other, specify (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Abdominal infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Anorectal infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Bronchial infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Catheter related infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 2 (3) | 6 (6)
Endocarditis infective (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Enterocolitis infectious (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 3 (3)
Hepatic infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Infections and infestations - Other, specify (Infections and infestations) | 5 (6) | 0 (0) | 0 (0) | 2 (2) | 6 (22) | 5 (9) | 23 (43)
Lung infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 3 (4) | 1 (1) | 1 (1)
Mucosal infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Peritoneal infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 1 (1) | 11 (14)
Skin infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Small intestine infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Soft tissue infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Tracheitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Upper respiratory infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 3 (3)
Wound infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Injury, poisoning and procedural complications - Other, specify (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Vascular access complication (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Activated partial thromboplastin time prolonged (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 3 (12) | 1 (4) | 10 (16)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (2) | 1 (4) | 8 (9)
Blood bilirubin increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 2 (2)
Creatinine increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Fibrinogen decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
GGT increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Investigations - Other, specify (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lipase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Lymphocyte count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (2) | 1 (2)
Neutrophil count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (2) | 2 (3) | 7 (10)
Platelet count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 3 (6)
Weight loss (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
White blood cell decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (2) | 2 (3) | 2 (5)
Acidosis (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Anorexia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 2 (2) | 6 (9)
Hyperglycemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypernatremia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 1 (1)
Hypertriglyceridemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypoalbuminemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 5 (6)
Hypocalcemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Hypoglycemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 3 (4)
Hypokalemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (3) | 1 (1) | 6 (6)
Hyponatremia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypophosphatemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Treatment related secondary malignancy (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abducens nerve disorder (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cognitive disturbance (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Depressed level of consciousness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Encephalopathy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Oculomotor nerve disorder (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Seizure (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 2 (2)
Stroke (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Psychiatric disorders - Other, specify (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Adult respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Apnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 4 (4)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 4 (5)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3)
Skin ulceration (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 3 (3)
Surgical and medical procedures - Other, specify (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 1 (1) | 5 (5)
Thromboembolic event (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Visceral arterial ischemia (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Induction (All Patients) (N=210) | Post Induction (Follow-up Only) (N=12) | Arm A (Standard Risk MLL-G) (N=60) | Arm B (IR/HR MLL-R Chemotherapy) (N=54) | Arm C (Safety/ Dose Level 1) (N=11) | Arm C (Safety/ Dose Level 2) (N=11) | Arm C (Efficacy/ Dose Level 2) (N=56)
Anemia (Blood and lymphatic system disorders) | 4 (4) | 0 (0) | 4 (7) | 4 (7) | 1 (2) | 1 (1) | 5 (7)
Blood and lymphatic system disorders - Other, specify (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Febrile neutropenia (Blood and lymphatic system disorders) | 31 (32) | 0 (0) | 34 (58) | 32 (69) | 6 (9) | 4 (13) | 26 (40)
Leukocytosis (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cardiac arrest (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cardiac disorders - Other, specify (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Myocarditis (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Sinus tachycardia (Cardiac disorders) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Blurred vision (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Eye disorders - Other, specify (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 1 (1) | 0 (0)
Anal mucositis (Gastrointestinal disorders) | 3 (3) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 2 (2)
Anal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Colitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 1 (1) | 1 (1) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 15 (16) | 0 (0) | 15 (21) | 14 (24) | 2 (5) | 1 (1) | 16 (28)
Dysphagia (Gastrointestinal disorders) | 3 (3) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Enterocolitis (Gastrointestinal disorders) | 2 (2) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Esophagitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastric hemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastritis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastrointestinal disorders - Other, specify (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 1 (1)
Mucositis oral (Gastrointestinal disorders) | 13 (14) | 0 (0) | 35 (46) | 24 (29) | 6 (9) | 5 (10) | 24 (30)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 3 (3) | 0 (0) | 1 (1)
Oral hemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Oral pain (Gastrointestinal disorders) | 2 (2) | 0 (0) | 2 (2) | 4 (4) | 1 (1) | 0 (0) | 1 (1)
Rectal mucositis (Gastrointestinal disorders) | 3 (3) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Small intestinal mucositis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 4 (4) | 0 (0) | 2 (3) | 6 (6) | 0 (0) | 0 (0) | 4 (4)
Death NOS (General disorders) | 0 (0) | 3 (3) | 0 (0) | 10 (10) | 3 (3) | 1 (1) | 3 (3)
Edema face (General disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Fatigue (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Fever (General disorders) | 2 (3) | 0 (0) | 9 (12) | 6 (7) | 2 (2) | 2 (3) | 2 (2)
General disorders and administration site conditions - Other, specify (General disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Hypothermia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Infusion related reaction (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Irritability (General disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 1 (2)
Multi-organ failure (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pain (General disorders) | 3 (3) | 0 (0) | 2 (2) | 2 (3) | 1 (1) | 0 (0) | 3 (3)
Hepatic failure (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Allergic reaction (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Anaphylaxis (Immune system disorders) | 1 (1) | 0 (0) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Immune system disorders - Other, specify (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Anorectal infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Bladder infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 1 (2)
Bronchial infection (Infections and infestations) | 2 (3) | 0 (0) | 3 (3) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Catheter related infection (Infections and infestations) | 5 (6) | 0 (0) | 13 (20) | 12 (21) | 3 (4) | 1 (3) | 8 (10)
Endocarditis infective (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3)
Enterocolitis infectious (Infections and infestations) | 4 (4) | 0 (0) | 3 (3) | 7 (8) | 0 (0) | 0 (0) | 1 (1)
Infections and infestations - Other, specify (Infections and infestations) | 52 (66) | 0 (0) | 32 (66) | 36 (116) | 4 (18) | 8 (11) | 19 (39)
Lung infection (Infections and infestations) | 4 (4) | 0 (0) | 5 (5) | 7 (11) | 1 (1) | 1 (1) | 5 (6)
Meningitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Mucosal infection (Infections and infestations) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Otitis media (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 1 (2) | 4 (5)
Paronychia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Penile infection (Infections and infestations) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rash pustular (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Scrotal infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 7 (7) | 0 (0) | 2 (2) | 10 (15) | 1 (1) | 0 (0) | 5 (7)
Sinusitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 2 (2) | 0 (0) | 0 (0)
Skin infection (Infections and infestations) | 3 (3) | 0 (0) | 7 (8) | 7 (9) | 2 (2) | 3 (4) | 1 (2)
Small intestine infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Soft tissue infection (Infections and infestations) | 1 (1) | 0 (0) | 3 (4) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Upper respiratory infection (Infections and infestations) | 6 (6) | 0 (0) | 7 (9) | 10 (15) | 0 (0) | 1 (1) | 6 (6)
Urinary tract infection (Infections and infestations) | 6 (6) | 0 (0) | 7 (9) | 21 (30) | 1 (2) | 3 (4) | 13 (14)
Vulval infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Wound infection (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Intraoperative hemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vascular access complication (Injury, poisoning and procedural complications) | 5 (5) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Wound complication (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Activated partial thromboplastin time prolonged (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Alanine aminotransferase increased (Investigations) | 24 (24) | 0 (0) | 42 (94) | 35 (84) | 8 (32) | 7 (12) | 30 (57)
Alkaline phosphatase increased (Investigations) | 0 (0) | 0 (0) | 4 (4) | 0 (0) | 1 (1) | 1 (1) | 1 (2)
Aspartate aminotransferase increased (Investigations) | 15 (15) | 0 (0) | 34 (52) | 28 (59) | 5 (11) | 4 (5) | 21 (31)
Blood bilirubin increased (Investigations) | 2 (3) | 0 (0) | 0 (0) | 4 (4) | 2 (3) | 0 (0) | 2 (2)
Creatinine increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
GGT increased (Investigations) | 3 (3) | 0 (0) | 3 (7) | 3 (4) | 2 (7) | 0 (0) | 3 (7)
Investigations - Other, specify (Investigations) | 3 (3) | 0 (0) | 1 (1) | 1 (4) | 0 (0) | 0 (0) | 1 (1)
Lipase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lymphocyte count decreased (Investigations) | 2 (2) | 0 (0) | 3 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Neutrophil count decreased (Investigations) | 74 (76) | 0 (0) | 29 (62) | 26 (45) | 9 (15) | 5 (8) | 26 (48)
Platelet count decreased (Investigations) | 9 (9) | 0 (0) | 9 (13) | 16 (24) | 4 (8) | 3 (5) | 12 (18)
Urine output decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Weight gain (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Weight loss (Investigations) | 3 (3) | 0 (0) | 4 (9) | 7 (12) | 0 (0) | 1 (1) | 0 (0)
White blood cell decreased (Investigations) | 6 (6) | 0 (0) | 14 (19) | 9 (13) | 2 (5) | 1 (1) | 8 (16)
Acidosis (Metabolism and nutrition disorders) | 4 (4) | 0 (0) | 1 (1) | 2 (3) | 1 (2) | 0 (0) | 0 (0)
Anorexia (Metabolism and nutrition disorders) | 18 (18) | 0 (0) | 13 (28) | 15 (31) | 2 (2) | 2 (5) | 9 (29)
Dehydration (Metabolism and nutrition disorders) | 4 (4) | 0 (0) | 8 (10) | 9 (16) | 1 (1) | 0 (0) | 5 (5)
Hypercalcemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hyperglycemia (Metabolism and nutrition disorders) | 19 (19) | 0 (0) | 4 (5) | 9 (17) | 3 (3) | 2 (2) | 7 (8)
Hyperkalemia (Metabolism and nutrition disorders) | 6 (6) | 0 (0) | 1 (1) | 3 (4) | 2 (2) | 0 (0) | 2 (2)
Hypernatremia (Metabolism and nutrition disorders) | 3 (3) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 2 (2)
Hypertriglyceridemia (Metabolism and nutrition disorders) | 3 (3) | 0 (0) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 2 (2)
Hypoalbuminemia (Metabolism and nutrition disorders) | 15 (15) | 0 (0) | 3 (3) | 5 (6) | 1 (1) | 0 (0) | 5 (6)
Hypocalcemia (Metabolism and nutrition disorders) | 29 (29) | 0 (0) | 5 (6) | 3 (5) | 0 (0) | 3 (3) | 5 (6)
Hypoglycemia (Metabolism and nutrition disorders) | 5 (5) | 0 (0) | 4 (6) | 2 (2) | 3 (5) | 0 (0) | 7 (8)
Hypokalemia (Metabolism and nutrition disorders) | 35 (36) | 0 (0) | 20 (37) | 14 (41) | 6 (16) | 3 (4) | 22 (37)
Hypomagnesemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (3)
Hyponatremia (Metabolism and nutrition disorders) | 14 (14) | 0 (0) | 5 (8) | 8 (9) | 2 (3) | 1 (1) | 2 (3)
Hypophosphatemia (Metabolism and nutrition disorders) | 5 (5) | 0 (0) | 2 (3) | 2 (2) | 3 (4) | 0 (0) | 3 (3)
Metabolism and nutrition disorders - Other, specify (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Muscle weakness trunk (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Leukemia secondary to oncology chemotherapy (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other, specify (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 4 (4) | 1 (1) | 1 (1) | 1 (1)
Encephalopathy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Intracranial hemorrhage (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nervous system disorders - Other, specify (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Peripheral motor neuropathy (Nervous system disorders) | 0 (0) | 0 (0) | 1 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Peripheral sensory neuropathy (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (3)
Insomnia (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hematuria (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Renal and urinary disorders - Other, specify (Renal and urinary disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Penile pain (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Adult respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Bronchopulmonary hemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 6 (6) | 0 (0) | 4 (8) | 3 (5) | 0 (0) | 1 (1) | 4 (4)
Laryngeal mucositis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pharyngeal mucositis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 1 (1) | 3 (3) | 0 (0) | 0 (0) | 1 (1)
Respiratory, thoracic and mediastinal disorders - Other, specify (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 4 (7) | 0 (0) | 0 (0) | 1 (1)
Sinus disorder (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Stridor (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Erythema multiforme (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pain of skin (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Periorbital edema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 4 (4) | 0 (0) | 3 (4) | 4 (6) | 0 (0) | 0 (0) | 1 (1)
Skin induration (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Skin ulceration (Skin and subcutaneous tissue disorders) | 12 (12) | 0 (0) | 5 (5) | 3 (3) | 0 (0) | 0 (0) | 8 (10)
Surgical and medical procedures - Other, specify (Surgical and medical procedures) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 25 (25) | 0 (0) | 1 (1) | 5 (8) | 0 (0) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 4 (4) | 0 (0) | 1 (2) | 5 (5) | 2 (3) | 1 (1) | 4 (4)
Thromboembolic event (Vascular disorders) | 2 (2) | 0 (0) | 0 (0) | 3 (3) | 1 (1) | 0 (0) | 1 (1)
Vascular disorders - Other, specify (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)

LIMITATIONS AND CAVEATS:
Data was and never will be collected for Outcome Measure #4, 5, 12, and 13.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Must obtain sponsor approval.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2013-04-05): https://cdn.clinicaltrials.gov/large-docs/93/NCT00557193/Prot_SAP_000.pdf